CLINICAL TRIAL: NCT02154620
Title: Dorsally Displaced Distal Radius Fractures in Patients Over 70 Years - Volar Plate or Plaster - A Prospective Randomized Trial
Brief Title: Distal Radius Fractures in Patients Over 70 Years - Volar Plate or Plaster
Acronym: 70
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sari Ponzer, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70
Record Dates: First submitted 2014-05-02; First posted 2014-06-03 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture; wrist fracture; volar plate; surgical treatment; plaster immobilisation
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plaster cast (No Intervention): The patient will be treated in a dorsal plaster cast for 4 weeks following the injury to the wrist
- Volar plate (Experimental): The patient will undergo surgery to the injured wrist with a Synthes Two-column plate (TCP) with a volar approach. Cast will be worn 2 weeks after surgery.
  Interventions: Procedure: Volar plate; Device: Synthes TCP volar plate

INTERVENTIONS:
Procedure: Volar plate — An anatomically countoured volar plate is implanted through a Henry's incision.
  Other Names: Synthes TCP volar plate for distal radius
  Arms: Volar plate
Device: Synthes TCP volar plate
  Arms: Volar plate

SUMMARY:
Distal radius fractures with dorsal dislocation among patients 70 years or older are randomized to conservative treatment with plaster or internal fixation with a volar plate. Thereafter they are followed at 2 weeks, 5 weeks, 3 months and 12 months with x-ray, functional scores and clinical examination.

An additional follow up at three years with X-ray, functional scores and clinical outcome will be conducted after a new written consent of continued participation in the study.

A health economy analysis will be preformed at 1, and 3 years for the participants with complete EQ5D.

ELIGIBILITY:
Inclusion Criteria:

* Dorsally displaced, 20 degrees or from a plane perpendicular do the diaphyseal axis, fracture.
* Low energy injury
* Patient 70 years old or older
* 72 hours or less since injury at time of diagnosis
* Patient registered in the Stockholm region
* Patient understands spoken and written swedish

Exclusion Criteria:

* Intraarticular displacement in radiocarpal joint of more than 1 mm
* Ulna fractured proximal to the base of the styloid process of ulna
* Earlier unilateral functional impairment of hand/wrist
* Injury to tendon, nerve or skin besides the fracture
* Rheumatoid arthritis or other severe systemic joint disease
* Severe psychiatric disorder, ongoing drug abuse or dementia (Pfeiffer score 5 points or less)
* Besides the wrist fracture also other big injuries, for example fracture of hip, shoulder or ankle
* Medical illness that makes general anesthesia impossible

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Patient related wrist evaluation (PRWE) | 52 weeks

SECONDARY OUTCOMES:
Patient related wrist evaluation (PRWE) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Enocson, M.D, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Orthopaedics, Stockholm South Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Sudow H, Severin S, Wilcke M, Saving J, Skoldenberg O, Navarro CM. Non-operative treatment or volar locking plate fixation for dorsally displaced distal radius fractures in patients over 70 years - a three year follow-up of a randomized controlled trial. BMC Musculoskelet Disord. 2022 May 12;23(1):447. doi: 10.1186/s12891-022-05394-7. PMID 35549696